CLINICAL TRIAL: NCT01817894
Title: Treatment With Topical Eflornithin After Laser Treatment in Women With Facial Hirsutism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Elisabeth Taudorf, MD PhD student, Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H-2-2011-139
Record Dates: First submitted 2013-02-14; First posted 2013-03-26 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Hirsutism
Keywords: Unwanted facial hair growth
MeSH Terms: conditions — Hirsutism | interventions — Eflornithine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- split-face eflornithin vs. no treatment (Other): Eflornithine cream 11.5 W/W% applied twice daily to one side of the face for six months
  Interventions: Drug: Eflornithine cream 11.5 w/w %

INTERVENTIONS:
Drug: Eflornithine cream 11.5 w/w % — Split face intervention with application of Eflornithine cream 11.5 w/w % versus no treatment for six months
  Other Names: Vaniqa

SUMMARY:
Split-face investigation of the efficacy of applying Eflornithin cream twice daily for six months after a period with six laser treatments for hair removal.

DETAILED DESCRIPTION:
Background: Unwanted facial hair growth is a serious problem for 5-15% of all women winch affects their quality of life. In Denmark patients are offered six laser treatments covered by the public health insurance. There is a lack of good follow-up treatments to this regime that can extent the efficacy of the laser treatment. Eflornithin cream is an approved treatment for reduction of facial hair growth which has proved to give an additional efficiency when used in combination with laser treatments.The efficacy when used after laser hair removal is not known.

Aim: To investigate whether an extended efficacy of laser hair removal can be achieved with application of Eflornithin cream twice daily for six months after completion of laser treatments.

Method: in a split-face trial to apply Eflornithin cream twice daily for six months. Outcome measures are investigator evaluation, blinded on-site evaluation, patient's assessment score and clinical photos.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* habile, understands Danish
* moderate to severe hirsutism prior to laser treatments
* succeeded minimum five laser treatments
* intact skin with no severe adverse events to laser treatments
* record of current medication and androgen hormone blood profile available
* Use of safe anti-conception (fertile women)

Exclusion Criteria:

* Pregnant or lactating
* allergy toward the content of Eflornithin cream
* Concomitant use of immunosuppressive therapy
* Dementia, psychiatric disease, alcoholic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
blinded photo-evaluation of change in facial hirsutism by hair count in a standardized square field | baseline, 1, 3 and 6 months

SECONDARY OUTCOMES:
Doctors blinded on-site evaluation of efficacy | Baseline, 1, 3 and 6 months
  Based on a four-point scale used on both sides of the face separately:
  * no effect
  * small effect (clearly visible hairs on evaluated side)
  * large effect (minimal hair on evaluated side)
  * significant effect (none or next to no hair on evaluated side)
Patient's overall satisfaction | Baseline, 1, 3 and 6 months
  Based on a VAS scale (0-10)
Patient's assessment of efficacy | Baseline, 1, 3 and 6 months
  Based on a four-point scale used on both sides of the face separately:
  * no effect
  * small effect (clearly visible hairs on evaluated side)
  * large effect (minimal hair on evaluated side)
  * significant effect (none or next to no hair on evaluated side)
Patient's assessment of adverse events | Baseline, 1, 3 and 6 months
  Five common side-effects (acne, rash, erythema, changes in pigment, stinging or burning sensation) are evaluated based on a four-point scale:
  1. none
  2. mild
  3. moderate
  4. severe Other observed side effects will also be registered and rated
Doctor's on-site blinded assessment of adverse events | Baseline, 1,3 and 6 months
  Five common side-effects (acne, rash, erythema, changes in pigment, stinging or burning sensation) are evaluated based on a four-point scale:
  1. none
  2. mild
  3. moderate
  4. severe Other observed side effects will also be registered and rated
Patient's overall impression of efficacy | Baseline, 1,3 and 6 months
  Assessment of the patients impression of difference between two sides of the face on a four-point scale:
  1. No difference
  2. little difference
  3. large difference
  4. significant difference, complete or almost complete clearance of hair on treated side.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth H Taudorf, MD, Principal Investigator — BispbejergH
Locations (1):
- Dermatological Dep Bispebjerg Hospital, Copenhagen NV, Copenhagen, Denmark